CLINICAL TRIAL: NCT07346183
Title: CommunityRx-Dementia + Peer Navigation (CRxDpeer): A Real-World Implementation and Effectiveness Study of an IT-Based Social Care Intervention
Brief Title: CommunityRx-Dementia + Peer Navigation (CRxDpeer)
Acronym: CRxDpeer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB25-1341; R01AG091308 (NIH)
Record Dates: First submitted 2026-01-14; First posted 2026-01-16 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer s Disease; Dementia; Caregiver; Loneliness; Health-Related Social Needs; Social Care; Healthcare Utilization; End of Life Care; Caregiver Burden; Anxiety; Stress; Depression; Self-Efficacy; Peer Support; Implementation Science; Advance Care Planning
Keywords: resource navigation; peer navigator; peer mentor; social care; dementia caregiver
MeSH Terms: conditions — Dementia; Caregiver Burden; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Cases will receive the CRxDpeer intervention plus usual care. Controls will not receive the intervention, but will receive the usual standard of care.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-Blind randomized controlled trial where the data collectors are blinded to the condition to which the subject has been assigned. The subject is also blinded to the condition they are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cases (Experimental): Usual care + CommunityRx-Dpeer
  Interventions: Other: CommunityRx-Dpeer
- Control (No Intervention): Usual Standard Care

INTERVENTIONS:
Other: CommunityRx-Dpeer — Essential components of the CRxDpeer intervention include: (1) focused education about common social (e.g. food, housing, transportation) and, specifically, caregiving needs (e.g. caregiver education, stress management, End of Life/Advance Care Planning (EOL/ACP)) and related resources, (2) activation of community resources through delivery of and coaching on use of a personalized local referral list (a "HealtheRx") and (3) boosting through a series of automated proactive text messages and ongoing resource navigational support by text/phone/email/video for utilizing resources. This intervention will be delivered by a peer mentor who is experienced in dementia caregiving and trained to provide 1:1 peer mentorship and resource navigation to dementia caregivers.
  Other Names: CRxDpeer
  Arms: Cases

SUMMARY:
The CRxDpeer intervention, delivered by a trained peer navigator, in practice called a "peer mentor", includes three evidence-based components: (a) focused education about common social (e.g., food and housing insecurity) and caregiving (e.g., respite and end of life care) needs, (b) activation of personalized community resource information for social and caregiving needs through delivery of a resource list (HealtheRx) at the baseline encounter and coaching on how to communicate with service providers, coordinate services and manage social support (e.g., connect with their peer navigator, reach out to friends or relatives for support, identify support groups, etc.) and (c) ongoing navigation-focused support meant to boost the baseline intervention, including a series of proactive text messages over 12 months. During this time, the subject can respond to and communicate with the peer navigator for ongoing support.

DETAILED DESCRIPTION:
In 2022, more than 11 million Americans, half of whom were 50 or older, provided more than 18 billion hours of unpaid care for people with dementia. Many caregivers have no formal training and limited support. The White House, along with the Alzheimer's Association, the National Institute on Aging and others, is calling for urgent attention to the health and well-being of the fast-growing population of dementia caregivers, with heightened concern for caregivers living in historically marginalized communities. Scalable, evidence-based, solutions leveraging existing assets are urgently needed to meaningfully reach all caregivers. Our approach to addressing these unmet needs, CommunityRxDpeer, is an information technology-based, low-intensity, health system-initiated community resource navigation intervention delivered to caregivers by peer caregiver navigators remotely over time. Essential components include education about common social, including caregiving needs, activation of personalized community resource information and ongoing navigation-focused support. The CRxDpeer intervention components are informed by evidence-based "processes" identified in the Grey et al. Self- and Family Management Framework that are known to promote desirable health outcomes among people living or caring for others with chronic health conditions, including dementia. Prior CommunityRx trials have successfully deployed community members, clinicians and researchers to deliver the intervention in real-world and research settings with positive outcomes in a wide-range of populations. In this pragmatic trial, experienced and willing dementia caregivers from the CRxDementia cohort (2020-24) will be recruited and trained as peer navigators to deliver CRxDpeer. Using a hybrid effectiveness implementation design with a double-blind RCT, we will evaluate the effectiveness of CRxDpeer versus usual care on caregiver health and well-being, healthcare utilization and social care outcomes. In parallel, we will evaluate the adoption, fidelity and cost of CRxDpeer and, using mixed methods, characterize perceived mechanisms of impact on caregivers delivering and receiving CRxDpeer. The specific objectives are to demonstrate that CRxDpeer can be delivered in the real world with fidelity and to assess the effectiveness of this approach on important outcomes. Resource referral and peer support IT platforms deployed for intervention delivery are already in commercial use, paving a viable path to replication and scale as a stand-alone or adjunct to other caregiver interventions, like the Center for Medicare & Medicaid Guiding an Improved Dementia Experience (GUIDE) Model test, which aims to enable people with dementia to age at home by supporting family caregivers with education and resources. CRxDpeer has the potential to improve the health and well-being of millions of dementia caregivers and their care recipients by meaningfully connecting them to vital social and caregiving resources and creating opportunity for willing and experienced caregivers to support with others.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as a caregiver of a home-dwelling person with Alzheimer's disease or related dementias (ADRD)
* Resides in the target geographic region of the study
* Has access to a cell phone and agrees to receive text messages from the study
* Has an email address that they can receive emails from
* Individuals under the age of 18 who are emancipated minors in the state of Illinois and a caregiver of a person with dementia

Exclusion Criteria:

* Minors who are not emancipated in the state of Illinois.
* Previously participated in the intervention arm of the CommunityRx-Dementia clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Caregiver loneliness at 6 months | 6 months
  Loneliness is measured using the 3-item UCLA Loneliness Scale (Hughes et al. 2004). Responses to each of the items are scored 1= "Hardly ever", 2= "Some of the time", or 3= "Often". A total score is generated by summing the individual items, with a possible range of 3-9 and higher scores = greater loneliness.
Caregiver's self-efficacy for finding end of life/advance care planning resources for the person with dementia at 12 months | 12 months
  Self-efficacy is measured using a single item question developed for this study: "How confident are you that you can find resources to help [name of care recipient] put into writing their medical wishes if they were very sick or near the end of their life?". Responses are measured on a 4-point scale of 1="Not at all confident", 2="Not very confident", 3="Somewhat confident", or 4="Completely confident" [higher score = greater self-efficacy].

IPD SHARING:
Plan to Share IPD: Undecided
In the interval since submission of our funding application, artificial intelligence (AI) capabilities and its application by the research community and the public more generally have evolved rapidly. In this context, we are re-examining our data sharing plan to optimize for both sharing and protection of human subjects against a potentially higher risk of deductive disclosure. We do plan to share de-identified data, or limited datasets, with researchers under approved IRB protocols.

REFERENCES:
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506